CLINICAL TRIAL: NCT01867814
Title: Clinical Trial for Evaluation of Arterial and Plethysmographic Waveform Variations as Predictors of Hemodynamic Response to Pneumoperitoneum During Laparoscopic Surgery
Brief Title: Arterial and Plethysmographic Waveforms Variables as Predictors of Hemodynamic Response to Pneumoperitoneum
Acronym: SPV-PnP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMC-12-0133-CTIL
Record Dates: First submitted 2013-05-27; First posted 2013-06-04 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Pneumoperitoneum; Heart Output Disorder
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pneumoperitoneum (Experimental): Patients undergoing laparoscopic surgery
  Interventions: Procedure: Pneumoperitoneum

INTERVENTIONS:
Procedure: Pneumoperitoneum — Pneumoperitoneum 15 mmHg and 10 mmHg

SUMMARY:
Laparoscopic surgery is frequently associated with hemodynamic changes due to pneumoperitoneum (PnP). Those complex hemodynamic changes are difficult to predict and occasionally they require active therapeutic interventions or even interruption of the surgical procedure.

One of the main hemodynamic effects of PnP is a decrease in cardiac output due to reduction of venous return and cardiac preload. Although it has been shown repeatedly that waveform variables are good predictors of cardiac output response to volume loading, the prediction hemodynamic response to decrease of preload is more complex.

The investigators hypothesize that waveform variables will predict cardiac output changes resulting from PnP. Particularly, augmented values of waveform variables before PnP will be associated with a larger decrease of cardiac output after establishing PnP.

DETAILED DESCRIPTION:
* Goals of the study

  * To evaluate hemodynamic changes caused by pneumoperitoneum applied for laparoscopic surgery
* Endpoints

  * Blood Pressure: Systolic, Diastolic, Mean (SBP, DBP, MBP)
  * Heart Rate (HR)
  * Cardiac Output/Index (CO/CI)
  * Stroke Volume/Index (SV/SVI)
  * Systolic Pressure Variation (SPV)
  * Stroke Volume Variation (SVV)
  * Plethysmographic Waveform Variation (PWV)
* Inclusion criteria

  * The patients scheduled for elective laparoscopic partial hepatectomy, laparoscopic splenectomy, laparoscopic pancreatectomy - required of continuous direct blood pressure monitoring according to the type of surgery
  * The patients ASA (American Society of Anesthesiologists)class III-IV scheduled for elective laparoscopic colectomy and hemicolectomy - required of continuous direct blood pressure monitoring according to their medical condition
  * Pneumoperitoneum by needle application only
  * Normal sinus cardiac rhythm
* Exclusion criteria

  * Patients that didn't sign informed consent
  * Patients ASA class I-II scheduled for elective laparoscopic colectomy or hemicolectomy
  * Patients scheduled for elective laparoscopic cholecystectomy
  * Patients required of monitoring by pulmonary artery catheter during the surgery according to their medical condition
* Study course, measurements and analysis

  * All study participants will get an explanation and sign on informed consent at least one day prior to the day of surgery
  * All study participants will receive standard anesthesia care. All patients will anesthetized intravenously with Fentanyl 2-5 mcg/kg, Propofol 1-2 mg/kg and Rocuronium 0.6-1.0 mg/kg followed by endotracheal intubation. Positive pressure ventilation with tidal volume 8 mL/kg of ideal body weight and respiratory rate 8-12 bpm to achieve end-tidal carbon dioxide of 33-37 mmHg will be applied after intubation. Anesthesia will be maintained with inhalation of Isoflurane (end-expiratory concentration at least 1.2%) in air/O2 (FiO2=0.4). Intraoperative fluid management will include an initial bolus of crystalloid solution (lactated Ringer's solution) at a dose of 7 mL/kg. Arterial blood pressure will be measured continuously through a radial arterial catheter. Pulse oximetry photoplethysmography will be monitored by index finger probe on the same side. Cardiac output will monitored noninvasively by NICOM (Non-invasive cardiac output monitor) that calculates stroke volume variation (SVV) in addition to cardiac output/cardiac index and stroke volume/stroke index
  * The study procedure will begin after induction of anesthesia, preparation of the patient for surgery and insertion of the pneumoperitoneum insufflation device. The study procedure will last for 10-15 minutes and will be finished before actual intraperitoneal surgical manipulation begins
* Waveforms will be recorded from the patient monitor and values of NICOM will be noted at baseline before surgical manipulation, at PnP pressure=0 mmHg before gas insufflation but after insertion of peritoneal needle, and after PnP pressure reaches 15 mmHg (routine value for laparoscopic surgery). If after reaching PnP pressure of 15 mmHg CO will decrease by more than 20%, the PnP pressure will be reduced to 10 mmHg and recording of waveforms will be repeated after two minutes
* Standard hemodynamic parameters (heart rate, systolic and diastolic BP) and waveform variables (SPV, PWV) will be measured and calculated offline according to the records
* Parameters measured by NICOM (CO, CI, SV, SVI, SVV) will be noted at baseline (PnP pressure=0 mmHg), after PnP pressure reached 15 mmHg and after PnP pressure decreased till 10 mmHg (if necessary)

  * There will be no further follow up of the patients
  * We anticipate that there will be a significant number of patients with a reduction of CO by 20% or more after establishment of PnP of 15 mm Hg. We will perform comparisons between waveforms at baseline between those who decrease CO and those who do not. If there will be significant difference in variables at baseline there will be justification to perform ROC analysis to evaluate sensitivity and specificity of these variables to predict decrease in CO. In patients who will have a decrease in CO after PnP of 15 mm Hg we will compare the same variables to those that will be reached at PnP of 10 mmHg. These comparisons can help to understand the mechanisms of CO decrease during PnP
  * All of the analysis of the data will be performed after removing all identifying data

ELIGIBILITY:
Inclusion Criteria:

* The patients scheduled for elective laparoscopic partial hepatectomy, laparoscopic splenectomy, laparoscopic pancreatectomy - required of continuous direct blood pressure monitoring according to the type of surgery
* The patients ASA class III-IV scheduled for elective laparoscopic colectomy and hemicolectomy - required of continuous direct blood pressure monitoring according to their medical condition
* Pneumoperitoneum by needle application only
* Normal sinus cardiac rhythm

Exclusion Criteria:

* Patients that didn't sign informed consent
* Patients ASA class I-II scheduled for elective laparoscopic colectomy or hemicolectomy
* Patients scheduled for elective laparoscopic cholecystectomy
* Patients required of monitoring by pulmonary artery catheter during the surgery according to their medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Cardiac output/cardiac index | Change of intraabdominal pressure before and 2-5 min after pneumoperitoneum
  Cardiac output/cardiac index will be measured before applying of pneumoperitoneum, 2-5 min after applying of pneumoperitoneum with intraabdominal pressure of 15 mmHg and 2-5 min after decrease of intraabdominal pressure until 10 mmHg

SECONDARY OUTCOMES:
Systolic pressure variation (SPV)/Pulse pressure variation (PPV) | Change of intraabdominal pressure before and 2-5 min after pneumoperitoneum
  Systolic pressure variation/Pulse pressure variation will be measured before applying of pneumoperitoneum, 2-5 min after applying of pneumoperitoneum with intraabdominal pressure of 15 mmHg and 2-5 min after decrease of intraabdominal pressure until 10 mmHg

OTHER OUTCOMES:
Plethysmographic Waveform Variation (PWV) | Change of intraabdominal pressure before and 2-5 min after pneumoperitoneum
  Plethysmographic Waveform Variation will be measured before applying of pneumoperitoneum, 2-5 min after applying of pneumoperitoneum with intraabdominal pressure of 15 mmHg and 2-5 min after decrease of intraabdominal pressure until 10 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Pizov Reuven, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- The Lady Davis Carmel Medical Center, Haifa, Israel